CLINICAL TRIAL: NCT05586763
Title: Comparison of Efficacy of Metoclopramide , Promethazine and Prochloroperazine in the Treatment of Vertigo.
Acronym: BBPVOMSBAFH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Asma Salim Abdullah Al Buraiki, Comparison of Efficacy of Metoclopramide , promethazine and prochloroperazine in the treatment of Vertigo., Oman Medical Speciality Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Omsb1993
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-06

CONDITIONS: Peripheral Vertigo
Keywords: ED; vertigo; metoclopramide; promethazine; Prochlorperazine
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Intervention Model Description: A 3-arm multi-center, randomized, triple-blind, controlled study comparing three treatments for acute vertigo Arm I : IM Metoclopramid ( 10mg) Arm II : IM Promethazine (25mg) Arm III : IM prochloraperazine( 12.5mg)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each patient with vertigo symptoms will be registered in vertigo list after written consent taken. The ED doctor will take one paper from the vertigo list box and will write the case there including patient ID, date, age and symptoms. Assessment (VAS ) will be done in the pre- medication, post medication 60 mins post intervention medication. The medication will be provided blindly through the pharmacy. Any possible medication side effect and any possible further work up done for patient will be involved in each paper as ED doctor will put a tick near each point. Score will be written in papers as per patient evaluation of their symptoms grade from 1-10 in three different positions (supine, sitting and standing). The need for rescue medication ( betahisten or ondansetron ) will be recorded in the paper as well as the need of eply manuver as rescue. Principle investigator in each centers will be responsible to collect the papers for analysis by end of each weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metoclopramid (Active Comparator): IM Metoclopramid 10mg
  Interventions: Drug: Metoclopramid ( 10mg), IM promethazine (25mg) , IM prochloroperazine( 12.5mg)
- Promethazine (Active Comparator): IM Promethazine 25mg
  Interventions: Drug: Metoclopramid ( 10mg), IM promethazine (25mg) , IM prochloroperazine( 12.5mg)
- prochloraperazine (Active Comparator): IM prochloraperazine 12.5mg
  Interventions: Drug: Metoclopramid ( 10mg), IM promethazine (25mg) , IM prochloroperazine( 12.5mg)

INTERVENTIONS:
Drug: Metoclopramid ( 10mg), IM promethazine (25mg) , IM prochloroperazine( 12.5mg) — Each patient with vertigo symptoms will be registered in vertigo list after written consent taken. The ED doctor will take one paper from the vertigo list box and will write the case there including patient ID, date, age and symptoms. Assessment (VAS & EEV) will be done in the pre- medication 0 min, and at 60 mins posts anti-vertigo medication. The medication will be provided blindly through the pharmacy. Any possible medication side effect and any possible further work up done for patient will be involved in each paper as ED doctor will put a tick near each point. Score will be written in papers as per patient evaluation of their symptoms grade from 1-10. The need for rescue medication ( betahisten or ondansetron ) will be recorded in the paper or is need eply manuver. Principle investigator in each centre will be responsible to collect the papers for analysis by end of each weeks.
  Other Names: Metoclopramid ( 10mg), IM phenergan (25mg) , IM stemetil( 12.5mg)

SUMMARY:
Background: Vertigo as acute symptom seem to be one of most common presentation in ED, can be treated in ED with multiple medication . Objective: This study aimed to compare the therapeutic efficacy of metoclopramide, promethazine and prochloroperazine in patients presenting with signs and symptoms suggestive of acute peripheral vertigo to the ED . Methods: A 3-arm multi-center, randomized, triple-blind, controlled study comparing three treatments for acute vertigo in three medical centers : AlNahdha hospital Oman , Sohar Hospital Oman and AFH hospital Oman. Oman From February 2022 to August 2024.

DETAILED DESCRIPTION:
* Background Vertigo is one of most ED visit symptoms, It can be due to central or peripheral cause. The most frequent three reasons for vertigo are acute peripheral vestibulopathy (vestibular neuritis, labyrinthitis), Meniere's disease, and benign paroxysmal positional vertigo (BPPV). Usually ED doctors started with Epley maneuver for relief of symptoms and then started with medication.
* Objective:

This study aimed to compare the therapeutic efficacy of metoclopramide, promethazine and prochloroperazine in patients presenting with signs and symptoms suggestive of acute peripheral vertigo to the ED .

• Research methods: This will be done by assessing the Best medication can be used to treat peripheral vertigo with least side effect through Randomized triple blinded analysis will use 3 medications. All medications will be saved in similar syringe with white paper cover and labeled as A,B, C .The treating EM Doctor will prescribe medication as anti-vertigo then one of covered medication will be randomly taken among 3 medication groups. Target population will be all patient in age group (18-60) years visiting the emergency department at Al Nahdha hospital, AFH and Sohar hospital who complain of peripheral vertigo after assessment and excluding central cause. Ethical approval will be applied for through the OMSB (Ministry of health ethical committee)

ELIGIBILITY:
Inclusion Criteria:

* □ Acute peripheral vertigo with nausea or vomiting (vas, visual analog scale >5) during their emergency department episode of care for which the attending physician recommending antiemetic, onset with in 3 days .

  * Age( 18- 60).

Exclusion Criteria:

* • Age >60.

  * Any organic brain disease (Clear central cause; "malignancy with brain metastasis".)
  * History of epilepsy
  * Pregnancy.
  * Dementia, Parkinson's disease
  * Abnormal vital signs
  * Any known drug allergy to the study drugs
  * Undergoing chemotherapy or radiotherapy
  * Mechanical bowel obstruction or perforation, gastrointestinal bleeding
  * Inability to understand study explanation or outcome measures (any reason)
  * Patients who refused to participate study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
medication effectiveness in peripheral vertigo. | 1hr
  1. Compare the effects of IM metoclopramide or IM promethazine or IM prochloroperazine in three randomizing groups in the treatment of peripheral Vertigo in emergency setting using Visual Analogue Scale taken from visual vertigo analogue scale/adapted from Longridge et al.,2002. (Nausea and vertigo scores as measured by Visual Analogue Scale that include patient assessmet of his symptoms in view of vertigo/ nausea/ vomiting)

SECONDARY OUTCOMES:
The need of rescue medication/ appearing of side effects. | 0-1hr
  The need for more rescue medications to relive the symptoms or for any appearing side effect at the time frame of assessment for vertigo symptom/ side effects like extrapyramidal side effect.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Al Buraiki, MD, Principal Investigator — Oman Medical Speciality Board
Locations (1):
- Al Nahdha hospital, AFH and Sohar hospital, Muscat, Oman